CLINICAL TRIAL: NCT01497171
Title: Safety and Efficacy of Transvaginal Mesh Colposuspension for Anterior Vaginal Prolapse: the Elevate vs. Anterior Colporrhaphy Trial
Brief Title: The ELEGANT Trial: Elevate Transvaginal Mesh vs. Anterior Colporrhaphy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Early termination of study due to changes in funding.
Sponsor: Emanuel Trabuco (Other)
Collaborators: American Medical Systems (Industry)
Responsible Party: Sponsor-Investigator, Emanuel Trabuco, Assistant Professor of Obstetrics-Gynegology, Consultant-OB/Gyn Surgery, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-000247
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: Cystocele; Bladder prolapse; Anterior prolapse; Vaginal prolapse; Uterine prolapse; Urinary incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse; Cystocele; Uterine Prolapse; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elevate Mesh (Active Comparator): Elevate transvaginal mesh - surgical repair of prolapse
  Interventions: Procedure: Elevate Mesh
- Anterior Colporrhaphy (Active Comparator): Anterior colporrhaphy - surgical repair of prolapse
  Interventions: Procedure: Anterior Colporrhaphy

INTERVENTIONS:
Procedure: Elevate Mesh — Transvaginal mesh repair of anterior vaginal prolapse
  Arms: Elevate Mesh
Procedure: Anterior Colporrhaphy — Traditional suture repair of anterior vaginal prolapse
  Arms: Anterior Colporrhaphy

SUMMARY:
This study is designed to compare the safety and efficacy of a commercially available mesh kit used for surgical repair of anterior vaginal wall prolapse with traditional suture repair surgery.

DETAILED DESCRIPTION:
This is a multicenter, double blinded, randomized controlled trial, comparing Elevate® System with Interpro® Lite™, Anterior and Apical Prolapse Repair System (American Medical Systems) and Anterior Colporrhaphy (anterior suture repair) in women with symptomatic pelvic organ prolapse, who have opted to have surgical repair.

The goals of the study are to compare both efficacy and safety of the two procedures and to compare the surgical impact of mesh and suture repairs on vaginal function.

The principal investigator is from Mayo Clinic in Rochester, Minnesota. Mayo Clinic will serve as the data gathering and coordination site for this multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

* Women with symptomatic pelvic organ prolapse who opt for a vaginal repair
* Require both apical and anterior compartment repairs
* Willing to return for follow-up visit
* Understand and have signed informed consent to undergo randomization
* Need both an apical and anterior repair
* All trial participants who have a uterus will require a hysterectomy

Exclusion Criteria:

* Known or suspected vulvodynia
* Known or suspected interstitial cystitis
* History of chronic pelvic pain
* Current pregnancy
* Desire to maintain fertility
* History of reconstructive pelvic surgery with synthetic mesh
* History of radical pelvic surgery
* History of pelvic radiation therapy
* Currently undergoing treatment for a malignancy
* Medically poor candidates for surgery

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Trabuco, MD, Principal Investigator — Mayo Clinic
Locations (6):
- United States (5):
  - Kaiser-Permanente - North Valley, Roseville, California
  - Kaiser-Permanente - Santa Clara, Santa Clara, California
  - Stanford University School of Medicine, Stanford, California
  - Washington Hospital Center - MedStar Health, Washington D.C., District of Columbia
  - The Carl & Edyth Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
- St. Hedwig's Krankenhaus, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 women were enrolled at the German site (St. Hedwig's). No subjects were enrolled at the US sites.
Period: Overall Study
Arm/Group | Elevate Mesh | Anterior Colporrhaphy
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 5 women were enrolled at the German site (St. Hedwig's). No subjects were enrolled at the US sites.
Groups:
- Total: Total of all reporting groups
Arm/Group | Elevate Mesh | Anterior Colporrhaphy | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Comparison of the Proportion of Subjects in Each Group, Who Achieve Anatomic Success at 12 Month Follow-up.
Description: Anatomical success will be measured using a composite index including: lack of specific prolapse symptoms, no interval treatment and no observed prolapse beyond 1 cm from the hymen.
Time Frame: 12 months
Population: No analysis was done due to early termination of the study.
Arm/Group | Elevate Mesh | Anterior Colporrhaphy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Elevate Mesh | Anterior Colporrhaphy
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elevate Mesh (N=2) | Anterior Colporrhaphy (N=3)
Endometrial Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of study due to changes in funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No